CLINICAL TRIAL: NCT05701254
Title: Skeletal Effects of Type 1 Diabetes on Low-Trauma Fracture Risk
Status: Recruiting | Type: Observational
Sponsor: Creighton University (Other)
Responsible Party: Sponsor
Other Study IDs: 1425624-3
Record Dates: First submitted 2022-12-21; First posted 2023-01-27 (Actual); Last update posted 2024-09-25 (Actual); Status verified 2024-09

CONDITIONS: Type 1 Diabetes; Osteopenia; Bone Loss; Fractures, Bone
Keywords: Bone; Cortical Bone; Mechanical Strength
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Bone Diseases, Metabolic; Fractures, Bone

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Transilial bone biopsy samples will be retained and stored for possible future testing. Type 1 Diabetics will be matched to non-diabetics. All subjects undergo the bone biopsy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Type 1 Diabetics: All participants will complete 4 visits over 6-8 weeks. Visit 1 is a screening visit which includes a physical exam, a bone mineral density scan, a blood draw and an EKG. Visit 2 consists of dispensing the Tetracycline antibiotic required for the bone biopsy. Visit 3 is the bone biopsy and includes a blood draw. Visit 4 is to remove the stitches.
  Interventions: Procedure: Transilial bone biopsy
- Non-Type 1 Diabetics: All participants will complete 4 visits over 6-8 weeks. Visit 1 is a screening visit which includes a physical exam, a bone mineral density scan, a blood draw and an EKG. Visit 2 consists of dispensing the Tetracycline antibiotic required for the bone biopsy. Visit 3 is the bone biopsy and includes a blood draw. Visit 4 is to remove the stitches.
  Interventions: Procedure: Transilial bone biopsy

INTERVENTIONS:
Procedure: Transilial bone biopsy — The transiliac bone biopsy will be performed on each subject under local anesthesia, and conscious sedation. From one skin incision located ~2cm posterior and inferior to the anterior-superior pelvic spine on one side of the pelvis, the investigators will obtain two iliac bone specimens, each 7.5 mm in diameter, cylindrical in shape, and including both inner and outer cortices and the intervening trabecular bone.

SUMMARY:
Patients with Type 1 Diabetes Mellitus (T1DM) have a higher risk of low-trauma (osteoporotic) fracture that is 7-12 times higher than non-diabetics. The bone density of people with Type 1 Diabetes is higher at the time of fracture than in non-diabetics. This suggests the presence of underlying bone tissue mechanical defects. The potential benefits to participants would be knowledge gained about their bone density and the results of laboratory tests. On a wider scale, there may be general benefits to society because the knowledge gained from this study may help better understand the effects of diabetes on bone health

DETAILED DESCRIPTION:
The investigators will enroll 40 female, postmenopausal, patients with T1DM, fracturing or non-fracturing, who are age 50 and over, and have had diabetes for more than ten years. The investigators will perform 2 transiliac (hip bone) biopsies on each subject, one for mechanical testing, tissue analysis of AGEs, enzymatic crosslinks and bone tissue-bound water in cortical bone, and the other for histomorphometry and high-resolution 3D imaging in trabecular bone. A matched, non-diabetic, healthy control will be enrolled at the time each T1DM is enrolled.

ELIGIBILITY:
Inclusion Criteria:

Criteria for enrollment of female diabetics

1. No chronic disease diagnoses that may affect bone, as confirmed by the PI.
2. Normal clinical history, physical, and clinical laboratory exam (except for usual complications of a 10+-year diabetic, i.e., ~minimal neuropathy or retinopathy, known, but asymptomatic mild vascular disease, etc.)
3. Glomelular Filtration Rate (GFR) >45 ml/min (Renal Association lower limit for "mild" kidney failure).
4. Willingness to sign a consent form.
5. Willingness to undergo a transilial bone biopsy incision that yields 2 bone specimens.
6. No abnormalities in clinical blood chemistry measurements (small, age-related decreases in GFR, will be permitted).
7. Caucasian

Criteria for each non-diabetic subject, compared to their matched diabetic:

1. Dual-energy x-ray absorptiometry (DXA) measures (BMD, gm/cm) must be within +/- 15% in total hip.
2. Body mass index (BMI) must be within +/-10%.
3. Age must be within +/- 5 years.
4. Caucasian

Exclusion Criteria:

1. Women who have had Type 1 diabetes for less than 10 years.
2. Non-insulin dependent Type 1 diabetic.
3. Less than 50 years old.
4. Less than 5 years post menopausal.

Min Age: 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Males will not be recruited in order to avoid gender-based confounding effects in the data analysis.
Study Population: 40 female type 1 diabetics (both fracturing and non-fracturing) and 40 matched healthy female controls. The investigators will enroll an age-matched, healthy, non-diabetic, non-fracturing female control who is 5 years past the onset of menopause. All of our subjects, diabetics and controls, will be Caucasians, free of diagnoses other than diabetes, and all will have DXA T-scores at the femoral neck and/or total hip and/or lumbar spine between -1.0 and -2.5, (i.e. none will have T-scores in the DXA T-score range of osteoporosis).
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2019-06-18 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Compare cortical bone tissue levels of pentosidine (AGE), pyridinoline (normal enzymatic collagen crosslinks), and matrix-bound water between T1DM and controls. | 6-8 weeks
  For different advance glycation endproducts (AGEs), a) pentosidine (PEN), b) pyrinoline (Pyd), and c) tissue water (TW), will be measured using Raman spectroscopy technique on bone biopsy tissue obtained from study participants. Raman spectra will be obtained from the embedded block surfaces using a confocal Raman spectrometer (Renishaw InVia Qontor, www.renishaw.de). These spectra will be collected at the interstitial, cement lines, and actively bone forming osteons with evident fluorescent labels. A continuous laser beam with an excitation of 785 nm and power of 10 mW will be focused through a Raman microscope (Leica DM2700M), using the 50x objective, down to a micrometer-sized spot on the sample.
  1. Pentosidine (PEN) [ratio]. PEN (Pentosidine) from the integrated area ratio of bands 1495 (PEN) cm-1 / 1450 cm-1 (methylene side chains (CH2)).
  2. Pyrinoline (Pyd) [ratio]. The pyridinoline (Pyd; enzymatic trivalent collagen cross-link) content is calculated as the absorbance height

SECONDARY OUTCOMES:
Compare cortical bone tissue heterogeneity in nanoindentation measures of modulus and hardness between T1DM and controls. | 6- 8 weeks
  Bone tissue's hardness and modulus will be quantified by using nanoindentation technique. The nanoindentation is a mechanical/material strength testing technique. The technique has been used in bone tissue from bone biopsies.
  1. Hardness [GPa-giga-pascal-N/m2]
  2. Modulus [GPa-giga-pascal-N/m2]

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed Akhter, PhD, Principal Investigator — Creighton University Osteoporosis Research Center
Locations (1):
- Creighton University Osteoporosis Research Center, Omaha, Nebraska, United States